CLINICAL TRIAL: NCT03625609
Title: Sexaffectivity in Autistic Spectrum Disorder: Observed Behaviors and Referred Needs in Adolescence
Brief Title: Sexaffectivity in Autistic Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Jordi Torralbas Ortega, RN, Parc Taulí Hospital Universitari
Other Study IDs: 2018/509
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Autistic Disorders Spectrum; Sexual Behavior; Adolescent Development; Sexual Inadequacy
MeSH Terms: conditions — Child Development Disorders, Pervasive; Sexual Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The WHO defines sexual health as a state of physical, emotional, mental and social well-being, related to sexuality, not only the absence of illness, dysfunction or disability. To acquire and maintain adequate sexual health, the sexual rights of all people must be respected, protected and fully exercised.

People with Autism Spectrum Disorder (ASD) present difficulties in the development of social interaction skills, among other problems that directly affect their sexual health. The consolidated prejudices and social myths related to the sexual affectivity of people with ASD, and in general to people with intellectual diversity, have meant that they do not pay any attention to the sexual health of this group in the assessment of their needs.

Main objectives: to understand the experience lived by young people with ASD and their caregivers in relation to the affective needs during adolescence and to know the cognitive and behavioral expression of the affective dimension of adolescents with ASD.

Mixed simultaneous design: qualitative based on the phenomenological paradigm, in order to establish the perceived needs of young adults with ASD, their families and the professionals who attend them, with the realization of focus groups and in-depth interviews. The second quantitative part will be developed in adolescents (12-18 years) and their families, evaluating the habitual behaviors and difficulties of Interaction in the affective expression, by means of questionnaires and self-administered scales. It will be necessary to sign the Informed Consent by all the participants, with the specific acceptance of the project by the CEIC of the investigator's center.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with ASD. 12-18 years old

Exclusion Criteria:

* Non defined

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys and girls with ASD who want to participate in the collection of a scale with their families. Ages between 12 years old and 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-11 (Actual); Primary Completion 2020-02-11 (Estimated); Study Completion 2020-07-11 (Estimated)

PRIMARY OUTCOMES:
Sexual Behaivor Scale | 12-18 years old
  The measure utilized was developed specifically for this research - the Sexual Behaviour Scale (SBS; see Appendix) - and was based upon previous studies and the issues these studies identified (cf. Haracopos and Pedersen, 1992; Ruble and Dalrymple, 1993). The SBS examined parents' reports of their child's: (1) social behaviour; (2) privacy awareness; (3) sex education; and (4) sexual behaviour; as well as (5) parental concerns about outcomes for their child.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordi Torralbas Ortega, Sabadell, Barcelona, Spain